CLINICAL TRIAL: NCT03076827
Title: Comparison of Cortisol and Cytokines in Morning and Afternoon Surgerys According to Circadian Rhythm of Cortisol
Brief Title: Effects of Surgery Start Time on Postoperative Interleukin-6, Interleukin-8, and Cortisol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jae Jun Lee, associate professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chuncheon201701
Record Dates: First submitted 2017-01-30; First posted 2017-03-10 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Hemiarthroplasty; Arthroplasty, Replacement, Hip
MeSH Terms: interventions — Arthroplasty, Replacement, Hip; Hemiarthroplasty

STUDY DESIGN:
Intervention Model Description: Patients receiving total hip replacement or hip hemiarthroplasty are divided into two groups: the morning surgery group and the afternoon surgery group. After surgery, cortisol, IL-6, IL-8 and VAS were measured and compared.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group to begin surgery(total hip replacement or hip hemi-arthroplasty) in the morning
  Interventions: Procedure: Total hip replacement; Procedure: Hemi-arthroplasty
- Group P (Experimental): Group to begin surgery(total hip replacement or hip hemi-arthroplasty) in the afternoon
  Interventions: Procedure: Total hip replacement; Procedure: Hemi-arthroplasty

INTERVENTIONS:
Procedure: Total hip replacement — Total hip replacement starts in the morning in group A and starts in the afternoon in group P.
Procedure: Hemi-arthroplasty — Hemi-arthroplasty starts in the morning in group A and starts in the afternoon in group P.

SUMMARY:
Cortisol is a hormone that increases after trauma or surgery and has circadian rhythm. It has a form that is increased in the morning and decreased in the evening. The investigators expected to be influenced by circadian rhythm according to the time of operation, and compared morning and afternoon surgery.

DETAILED DESCRIPTION:
44 patients to undergo hip hemiarthroplasty or total hip replacement were divided to morning surgery group(Group A) and afternoon surgery group(Group P). All surgery was done by the same orthopedic surgeon. Anesthesia of Group A was started at 8 a.m. and Group P was at 12~2 p.m. Blood sampling was performed at 7:30 a.m., after induction of anesthesia, 6, 12, 24 and 48 hours after surgery in all patients of both groups. Cortisol, IL-6, and IL-8 was measured immediately after blood sampling. Visual analogue scale(VAS) was used to assess the degree of pain at before start of anesthesia, 6, 12, 24 and 48 hours after surgery. The postoperative hospital stay was calculated. Postoperative management was done by the same management team. Surgical wounds were treated at the same 24 hour intervals.

A sample size was calculated to differentiate between groups. Because difference of cortisol according to groups in ANOVA based on pilot study, the sample size was 20 patients per group. (Effect size f(v)= 0.5297047, α=0.05, 1-β=0.90) The investigators recruited total 44 patients to cover dropout 10%.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for hip hemiarthroplasty
* Patients scheduled for total hip replacement

Exclusion Criteria:

* Sleep disorder
* Mental disorder
* Psychiatric medication

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Cortisol level | within the first 2 days after surgery
  Cortisol levels over time

SECONDARY OUTCOMES:
Interleukin-6 | within the first 2 days after surgery
  Interleukin-6 levels over time
Interleukin-8 | within the first 2 days after surgery
  Interleukin-8 levels over time
Visual analogue scale | within the first 2 days after surgery
  pain scale over time
Post-operative hospital stay | Hospital day after surgery.
  Hospital day after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Jun Lee, M.D., Principal Investigator — Department of Anesthesiology and Pain medicine, Chuncheon Sacred Heart Hospital,

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Popma A, Doreleijers TA, Jansen LM, Van Goozen SH, Van Engeland H, Vermeiren R. The diurnal cortisol cycle in delinquent male adolescents and normal controls. Neuropsychopharmacology. 2007 Jul;32(7):1622-8. doi: 10.1038/sj.npp.1301289. Epub 2007 Jan 17. PMID 17228341
- [Derived] Kwon YS, Jang JS, Hwang SM, Tark H, Kim JH, Lee JJ. Effects of surgery start time on postoperative cortisol, inflammatory cytokines, and postoperative hospital day in hip surgery: Randomized controlled trial. Medicine (Baltimore). 2019 Jun;98(24):e15820. doi: 10.1097/MD.0000000000015820. PMID 31192911
- See also: Click here for more information about background of this study — https://www.ncbi.nlm.nih.gov/pubmed/?term=neuropsychipharmacology+2007+32++1622-1628